CLINICAL TRIAL: NCT04831853
Title: Comparison for Sensitivity and Tolerance of Self-swabbing and Conventional Nasopharyngeal Swabbing for SARS-CoV-2 Detection for Pain, Discomfort and Acceptability: a Randomized Controlled Non-inferiority Study
Brief Title: Self- Versus Conventional-swabbing for COVID-19 Screening (COVISWAB)
Acronym: COVISWAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2020 MOISSET 2; 2020-A02913-36 (Other: ANSM)
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: SARS-CoV-2; COVID-19; Nasopharyngeal swabbing; Self-swabbing; pain; Sensitivity
MeSH Terms: conditions — COVID-19; Pain; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized sequence of supervised self-swabbing and conventional swabbing for SARS-CoV-2 screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised self-swabbing followed by conventional swabbing (Experimental): the subjects will first benefit from a 5 minutes explanation on how to perform self-swabbing and will then performed the swabbing under the supervision of a trained healthcare professional
  Interventions: Other: nasopharyngeal swabbing procedure (self swabbing first)
- Conventional swabbing followed by supervised self-swabbing (Experimental): the subject will undergo conventional nasopharyngeal swabbing performed by a trained healthcare professional first.
  Interventions: Other: nasopharyngeal swabbing procedure (conventionnal swabbing first)

INTERVENTIONS:
Other: nasopharyngeal swabbing procedure (self swabbing first) — Patient realises the nasal swabbing himself first, then undergoes conventionnal swabbing
  Arms: Supervised self-swabbing followed by conventional swabbing
Other: nasopharyngeal swabbing procedure (conventionnal swabbing first) — patient undergoes conventionnal swabbing first then realises the nasal swabbing himself
  Arms: Conventional swabbing followed by supervised self-swabbing

SUMMARY:
Self-swabbing requires less personal protective equipment and could allow to test more people and even to do quick self-diagnosis if antigenic tests are available.

In a preliminary study on 190 medical students, the investigators have shown that self and conventional swabbing were identically well-accepted with equivalent level of pain and discomfort induced by swabbing. In a sub-group of this sample, the investigators have shown that the quality of the 2 sampling methods were equivalent.

The goal of this large study in the general population is to confirm these findings in an adequately powered study. Such results would allow to develop self-swabbing for large screening campaigns and eventually self-diagnosis using antigenic tests.

DETAILED DESCRIPTION:
All consecutive subjects coming to the 2 dedicated centers for COVID-19 screening in Clermont-Ferrand University hospital (one for medical students and one for the general population) will be asked to be included in the present study. They will be randomly assigned to either supervised self-swabbing followed by conventional swabbing led by a healthcare professional or the other way round.

All the subjects will have to complete a brief questionnaire including demographical characteristics (age, sex, height, weight, eye color), potential symptoms (asthenia, fever, anosmia…) anticipated pain and discomfort and previous nasopharyngeal swabbing experience. Pain, discomfort and overall acceptability of the procedure will be completed just after completion of the swabbing.

ELIGIBILITY:
Inclusion Criteria:

* Any subject coming for nasopharyngeal swabbing for SARS-CoV-2 screening
* Fluent in French (both oral and written)
* Able to give an eclaired consent

Exclusion Criteria:

* Contra-indication to nasopharyngeal swabbing
* Refusal to participate
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of self-swabbing compared to conventional swabbing concerning diagnosis sensitivity | 5 minutes after the end of the procedure of nasopharyngeal swabbing
  assessed using consistency of COVID-19 RT-PCR results for both sampling modalities (Self- swabbing versus conventional-swabbing). If non-inferiority is confirmed on this criterion, pain will be tested.

SECONDARY OUTCOMES:
Correlation between age, sex and swabbing-induced pain | 5 minutes after the end of the procedure
  Score on the pain numeric rating scale (0 to 10; higher scores meaning more pain)
Correlation between eye color and swabbing-induced pain | 5 minutes after the end of the procedure
  Eye-color self-reported by the subject on a validated 14 item scale and pain score on the numeric rating scale (NRS) (0 to 10; higher scores meaning more pain)
Correlation between eye color and swabbing-induced discomfort | 5 minutes after the end of the procedure
  Eye-color self-reported by the subject on a validated 14 item scale and discomfort score on numeric rating scale (0 to 10; higher scores meaning more discomfort)
Correlation between symptoms (fever, headache, asthenia, anosmia, agueusia, cough, dyspnea, muscle pain, sore throat, diarrhea) and swabbing-induced pain | 5 minutes after the end of the procedure
  symptoms self-reported by the subject and pain score on numeric rating scale (0 to 10; higher scores meaning more pain)
Correlation between body mass index and swabbing-induced pain | 5 minutes after the end of the procedure
  symptoms self-reported by the subject and pain score on numeric rating scale (0 to 10; higher scores meaning more pain)
Correlation between anticipated pain and actual pain | 5 minutes after the end of the procedure
  anticipated and actual pain self-reported on numeric rating scale (0 to 10; higher scores meaning more pain)
Correlation between anticipated discomfort and actual discomfort. | 5 minutes after the end of the procedure
  anticipated and actual discomfort self-reported on numeric rating scale (0 to 10; higher scores meaning more pain)
Richness assessment for respiratory cells | Day 0
  Ct value of beta-globin gene
Non-inferiority of self-swabbing compared to conventional swabbing concerning pain | 5 minutes after the end of the procedure of nasopharyngeal swabbing
  assessed using a Numerical Rating Scale (0 indicating no pain and 10 the worst imaginable pain). If non-inferiority is confirmed on this criterion, discomfort will be tested
Non-inferiority of self-swabbing compared to conventional swabbing concerning pain discomfort | 5 minutes after the end of the procedure of nasopharyngeal swabbing
  assessed using a Numerical Rating Scale (0 indicating no discomfort and 10 the worst imaginable discomfort). If non-inferiority is confirmed on this criterion, acceptability will be tested
Non-inferiority of self-swabbing compared to conventional swabbing concerning acceptability | 5 minutes after the end of the procedure of nasopharyngeal swabbing
  assessed using a Numerical Rating Scale (0 indicating that the procedure is not acceptable at all and 10 that the procedure is perfectly well accepted).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MOISSET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France